CLINICAL TRIAL: NCT03826732
Title: Guided Self-help Based on Acceptance and Commitment Therapy to Reduce Perceived Stress
Brief Title: Acceptance and Commitment Therapy (ACT) Self-help to Reduce Stress
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ata Ghaderi, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGFLDE
Record Dates: First submitted 2019-01-24; First posted 2019-02-01 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Randomization into active treatment versus a wait-list control group
Masking Description: Given the nature of the intervention, and self-report as a main strategy for outcome assessment, nor masking is possible or necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided self-help based on ACT (Experimental): Participants follow a self-help program and receive weekly support by trained facilitators
  Interventions: Behavioral: Guided self-help based on ACT
- Wait-list control (No Intervention): Participants are informed that they will receive the intervention after the 6-month follow-up assessment

INTERVENTIONS:
Behavioral: Guided self-help based on ACT — ACT-based self-help book and regular support by trained facilitators
  Arms: Guided self-help based on ACT

SUMMARY:
The efficacy of guided self-help based on acceptance and commitment therapy (ACT) to reduce subjective sense of stress will be investigated in a randomised controlled trial with two condition: 1) ACT-based self-help, and 2) Wait-list control. The outcome at the end of the treatment (week 10) and 6-month follow-up will be assessed. The wail-list condition will be offered ACT-based self-help after the post-assessment.

DETAILED DESCRIPTION:
The efficacy of guided self-help based on acceptance and commitment therapy (ACT) to reduce subjective sense of stress will be investigated in a randomised controlled trial with two condition: 1) ACT-based self-help, and 2) Wait-list control. The outcome at the end of the treatment and 6-month follow-up will be assessed. The wail-list condition will be offered ACT-based self-help after 10 weeks (i.e. when the post-assessment is completed). Inclusion criteria are: Adults with a score above 14 on the stress sub scale of the Depression, Anxiety, Stress Scale (DASS) at screening, a score below 10 on the Patient Health Questionnaire (PHQ-9), no indication of suicidality on the PHQ-9, and no ongoing psychotherapeutic interventions, and no previous work with the self-help manual that has been published as a self-help book.

A total of 140 participants will be recruited and randomised, using services on www.random.org. Informed consent will be obtained from all the participants ahead of screening. Participants will be asked to respond to the following questionnaires at pre-, post and follow-up assessments: Perceived Stress Scale-14 (PSS-14), General Anxiety Disorder-7 (GAD-7), Shirom Melamed Burnout Measure (SMBM), and Brunnsviken Brief Quality of Life Inventory (BBQ). Initially, they will also be asked to respond to the credibility/Expectancy Questionnaire (CEQ).

At the end of the intervention (week 10), participants will also be asked to respond to the Client Satisfaction Questionnaire (CSQ), and the Negative Effects Questionnaire (NEQ).

The following two scales will be used to study mediators: Acceptance and Action Questionnaire-2 (AAQ-2), and Attention Awareness Scale (MAAS), assess at pre-treatment, as well as at third and fifth week of treatment, at post-assessment (10 weeks later), and at the 6 months follow-up. A number of moderators, including demographics, will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* DASS score above 14
* PHQ-9 below 9

Exclusion Criteria:

* Any indications of suicidality
* Any indication of other psychiatric disorder in need of immediate attention/treatment
* Concurrent psychotherapy or other treatments for stress
* Previous work with the self-help book

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale-14 (PSS-14) | Pre-assessment, week 3 and 5 of intervention, post-assessment (week10), and 6 months follow-up
  The PSS-14 is measure of stress. Its total score ranges from 0-56. Lower values represent a better outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Pre- and post-assessment (10 weeks later) as well as 6 months follow-up
  The PHQ-9 provides a measure of depressive symptomatology. It ranges from 0-27. Lower values represent a better outcome
General Anxiety Disorder-7 (GAD-7) | Pre- and post-assessment (10 weeks later) as well as 6 months follow-up
  The GAD-7 is used to measure anxiety. It ranges from 0-21. Lower values represent a better outcome.
Brunnsviken Brief Quality of Life Inventory (BBQ) | Pre- and post-assessment (10 weeks later) as well as 6 months follow-up
  The BBQ is a Swedish measure of quality of life. It ranges from 0-96. Higher values represent a better outcome.
Shirom Melamed Burnout Measure (SMBM) | Pre- and post-assessment (10 weeks later) as well as 6 months follow-up
  The SMBM provides a measure of burn-out. It has three sub-scales: 1) physical exhaustion, 2) cognitive fatigue, and 3) emotional exhaustion. The subscales are combined to compute a total score by summing the mean of the subscales. Scale ranges from 3-15. Higher values represent a better outcome.
Acceptance and Action Questionnaire-2 (AAQ-2) | Pre-assessment, week 3 and 5 of intervention, post-assessment (week10), and 6 months follow-up
  To Measure psychological flexibility (mediator of change). It ranges from 7-49. Lower values represent a better outcome.
Mindful Attention Awareness Scale (MAAS) | Pre-assessment, week 3 and 5 of intervention, post-assessment (week10), and 6 months follow-up
  To measure mindfulness (potential mediator of change). The score is computed by the mean of the 15 items and the resulting scale ranges from 1-6. Higher values represent a better outcome.
Client Satisfaction Questionnaire (CSQ) | Post-assessment, and 6 month follow-up
  To measure satisfaction and dissatisfaction with the intervention. It ranges from 8-32. Higher values indicate higher satisfaction.
Negative Effects Questionnaire (NEQ) | Post-assessment, and 6 month follow-up
  To identify iatrogenic events. It ranges from 0-128. Lower values represent a better outcome (i.e. fewer negative effects from the intervention).

OTHER OUTCOMES:
Credibility/Expectancy Questionnaire (CEQ) | Pre-assessment
  To measure the perceived credibility of the intervention as well as expectations. It has two subscales; 1) expectancy, and 2) credibility. The individual items are first standardized and then summed up in each subscale. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ata Ghaderi, PhD, Principal Investigator — Professor
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data will be made available to other researchers upon request.
Supporting Information: ICF, Analytic Code